CLINICAL TRIAL: NCT05678192
Title: Optimization of Management Tactics for Postmenopausal Patients in Need of Menopausal Hormone Therapy, Taking Into Account the Effect on the Parameters of the Immune System
Brief Title: Effect of Menopausal Hormone Therapy on Immune System Parameters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-11/11.2021
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Last Period Not Earlier Than 6 Months Ago
Keywords: immune status; menopausal hormone therapy
MeSH Terms: interventions — Hormone Replacement Therapy

STUDY DESIGN:
Intervention Model Description: The cohort was divided into groups depending on the treatment regimen. Group 1 (n=20) received transdermal menopausal hormone therapy (MHT). Group 2 (n=20) received oral MHT.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdermal MHT (Other): The group includes women 45-59 years old, with menopausal symptoms. The choice of transdermal MHT was based on personal history (chronic diseases of the gastrointestinal tract, high blood pressure, etc.), family history (stroke, thromboembolism in relatives, etc.), and patient preferences. Used estradiol hemihydrate 0.6 mg 2 protective pumps. The progesterone component of MHT includes micronized progesterone 100 mg or 200 mg, depending on the MHT regimen (continuous or cyclic). Blood sampling to determine the immune status is carried out before the start of therapy after 3 months.
  Interventions: Drug: oral menopausal hormone therapy; Drug: transdermal menopausal hormone therapy
- Oral MHT (Other): The group includes women 45-59 years old, with menopausal symptoms. Examination before the appointment of MHT can be carried out according to clinical recommendations. The choice of transdermal MHT was based on the history (chronic diseases of the gastrointestinal tract, high blood pressure, etc.), family history (stroke, thromboembolism in relatives, etc.), the patient's preferences.Drugs used in this group include:
  Dydrogesterone 5 mg + Estradiol 1 mg or Dydrogesterone 10 mg + Estradiol 1 mg, depending on the MHT regimen. Blood sampling to determine the immune status is performed before the start of therapy and after 3 months
  Interventions: Drug: oral menopausal hormone therapy; Drug: transdermal menopausal hormone therapy

INTERVENTIONS:
Drug: oral menopausal hormone therapy — Dydrogesterone 10 mg + Estradiol 1 mg/Dydrogesterone 5 mg + Estradiol 1 mg
Drug: transdermal menopausal hormone therapy — Estradiol 1,5 mg + Progesterone 200 mg/Estradiol 1,5 mg + Progesterone 100 mg

SUMMARY:
The objective of the study is to evaluate the effect of menopausal hormone therapy on the parameters of the immune system. To do this, patients took blood to assess the immune status before the start of therapy and after 3 months.

An additional task is to assess the content of blood sex hormones before the start of therapy and after 3 months.

DETAILED DESCRIPTION:
A study of 60 perimenopausal and postmenopausal patients was included. The cohort was divided into groups depending on the treatment regimen.

Group 1 (n=20) received transdermal menopausal hormone therapy (MHT). Group 2 (n=20) received oral MHT.

ELIGIBILITY:
Inclusion Criteria:

* age from 45 to 59;
* phase of reproductive aging - perimenopause, postmenopause or surgical menopause (ovariectomy);
* indications for prescribing MHT

Exclusion Criteria:

1. Absolute contraindications to MHT:

   * Bleeding from the genital tract of unknown origin
   * Breast and endometrial cancer
   * Acute hepatitis
   * Acute deep vein thrombosis
   * Acute thromboembolism
   * Cutaneous porphyria
2. Obesity;
3. HIV infection and other congenital and acquired immunodeficiencies;
4. Systemic connective tissue diseases;
5. Oncological diseases in history;
6. History of chemotherapy and/or radiation therapy;
7. Autoimmune diseases;
8. Acute diseases and exacerbation of chronic diseases during the last 3 months;
9. Reception of immunomodulatory drugs during the last 3 months.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the severity of menopausal syndrome | 3 months
  The Green scale questionnaire was used initially and after 3 months against the background of menopausal hormone therapy. The questionnaire includes 21 questions from 0 to 3 points, where a lower score means a better result.
Changing the assessment of quality of life using the WHO Brief Questionnaire for Quality of Life (WHOQOL-BREF) | 3 months
  The WHO Brief Questionnaire for Quality of Life (WHOQOL-BREF) was used at baseline and 3 months later. The questionnaire includes 26 questions, from 1 to 5 points, where a higher score means a better result.

SECONDARY OUTCOMES:
Evaluation of the effect of therapy on the parameters of the immune status | 3 months
  Determination of blood parameters of immune status: the content cytotoxic T-lymphocytes (CD3+CD8+) in peripheral blood by flow cytometry in %. Literature reference values: 14,0-36,0%.
Evaluation of the effect of therapy on the parameters of the immune status | 3 months
  Determination of blood parameters of immune status: content of B-lymphocytes (CD3-CD19+HLA-DR+) in peripheral blood by flow cytometry in %. Literature reference values: 5,0-19,0%.
Evaluation of the effect of therapy on the parameters of the immune status | 3 months
  Determination of blood parameters of immune status: content of NK cells (CD3-CD56+CD16+) by flow cytometry in %. Literature reference values: 4,0-26,0%.
Evaluation of the effect of therapy on the parameters of the immune status | 3 months
  Determination of blood parameters of immune status: content of classical monocytes (CD14++CD16-) by flow cytometry in %. Literature reference values: 85,0-90,0%.
Evaluation of the effect of therapy on the parameters of the immune status | 3 months
  Determination of blood parameters of immune status: content of non-classical monocytes (CD14+CD16++) by flow cytometry in %. Literature reference values: 5,0-10,0%.
Evaluation of the effect of therapy on the parameters of the immune status | 3 months
  Determination of blood parameters of immune status: content of T-helper cells (CD3+CD4+) by flow cytometry in %. Literature reference values: 31,0-61,0%.

OTHER OUTCOMES:
Сhanges in the level of sex hormones against the background of MHT | 3 months
  Assessment of changes in the level of sex hormone in peripheral blood: follicle-stimulating hormone (IU/l). Reference values: 2.0-10.0 IU/l. Blood sampling is performed at baseline and after 3 months.
Сhanges in the level of sex hormones against the background of MHT | 3 months
  Assessment of changes in the level of sex hormone in peripheral blood: estradiol (pmol/l). Reference values: 150 - 450 pmol/l. Blood sampling is performed at baseline and after 3 months.
Сhanges in the level of sex hormones against the background of MHT | 3 months
  Assessment of changes in the level of sex hormone in peripheral blood: testosterone (nmol/l). Reference values: 0,52 - 2,5 nmol/l. Blood sampling is performed at baseline and after 3 months.
Assessing satisfaction with MHT using the Menopause symptoms treatment Satisfaction Questionnaire | 3 months
  The Menopause symptoms treatment Satisfaction Questionnaire is used after 3 months of MHT. The questionnaire includes 8 questions from 1 to 5 points from a very satisfactory result to a completely unsatisfactory one.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Averyanova, PhD, Principal Investigator — FSBI "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov" Ministry of Healthcare of the Russian Federation
Locations (1):
- Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare, Moscow, Russia